CLINICAL TRIAL: NCT01600573
Title: A Phase I/II Study of Pazopanib and Weekly Topotecan in Patients With Platinum-resistant or Intermediate-sensitive Recurrent Ovarian Cancer
Brief Title: Pazopanib and Weekly Topotecan in Patients Recurrent Ovarian Cancer (TOPAZ)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: JSehouli (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, JSehouli, Prof. Dr. Jalid Sehouli, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PazTo_2010
Record Dates: First submitted 2012-05-09; First posted 2012-05-17 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pazopanib plus weekly topotecan (Experimental): pazopanib in combination with weekly topotecan
  Interventions: Drug: pazopanib in combination with weekly topotecan

INTERVENTIONS:
Drug: pazopanib in combination with weekly topotecan — * Topotecan as an IV infusion over 30 minutes on days 1, 8, and 15 of a 28 day cycle and
  * Pazopanib orally once daily continuous dosing in the following dose levels:
  Phase I Trial:
  Dose level -I: Topotecan weekly 3mg/m2, Pazopanib 400 mg Dose level I: Topotecan weekly 4mg/m2, Pazopanib 400 mg Dose level II: Topotecan weekly 4mg/m2, Pazopanib 600 mg Dose level III: Topotecan weekly 4mg/m2, Pazopanib 800 mg
  Phase II Trial:
  Phase II will either use the MTD as determined in Phase I or a lower dose if deemed necessary.
  Other Names: pazopanib in combination with weekly topotean

SUMMARY:
This clinical trial shall clarify the efficacy and safety of pazopanib in combination with weekly topotecan in patients with platinum-resistant or intermediate platinum-sensitive recurrent epithelial ovarian cancer, fallopian and peritoneal carcinoma

DETAILED DESCRIPTION:
This study is a prospective single-arm, open-label, multicenter phase I/II trial. The phase I-trial is a dose-escalation trial to determine the maximum tolerated dose (MTD) of pazopanib in combination with weekly topotecan. The phase II-trial is a single arm open-label trial to further assess the safety and the efficacy of this combination of treatment.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* histologically confirmed diagnosis of epithelial ovarian cancer, primary peritoneal carcinoma or fallopian tube cancer
* platinum resistant (recurrence within 6 months of a platinum-containing regimen) or platinum refractory (progression during platinum treatment) or intermediate platinum-sensitive (recurrence within 12 months after a platinum-based primary therapy) disease
* no more than 2 prior treatment regimens for epithelial ovarian cancer
* Age more than 18 years
* ECOG of 0 or 1
* adequate organ function
* measurable disease or evaluable disease according to RECIST criteria
* able to swallow and retain oral medication
* life expectancy of at least 12 weeks
* non-childbearing potential or negative serum pregnancy test of women of childbearing potential and agrees to use adequate contraception for 14 days before exposure to investigational product, through the dosing period, and for at least 6 months after the last dose of investigational product. Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

Exclusion Criteria:

* prior malignancies; subject who have had another malignancy and have been disease-free for 5 years which effect progression free survival, or subject with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
* clinically significant gastrointestinal abnormalities that might interfere with oral dosing or that may increase the risk for gastrointestinal bleeding
* clinically significant gastrointestinal abnormalities that may affect absorption of investigational product
* Grade 3 or 4 diarrhoea
* Any unstable or serious concurrent condition (e.g., active infection requiring systemic therapy)
* poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg]
* Prolongation of corrected QT interval (QTc) >450 milliseconds using Bazett's formula
* History of any one or more of the following cardiovascular conditions within the past 6 months: Cardiac angioplasty or stenting; myocardial infarction; unstable angina; symptomatic peripheral vascular disease; coronary artery by-pass graft surgery
* Class III or IV congestive heart failure as defined by the New York Heart Association (NYHA)
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
* Macroscopic hematuria
* Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug
* Evidence of active bleeding or bleeding diathesis
* known endobronchial lesions and/or lesions infiltrating major pulmonary vessels and/or involvement of large pulmonary vessels by tumor
* prior major surgery or trauma within 14 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer
* Chemotherapy or radiation therapy or tumour embolization within 2 weeks prior to the first dose of study drug
* biological therapy, immunotherapy, hormonal therapy or treatment with an investigational agent within 14 days (for bevacizumab, 60 days) or 5 half-lives, whichever is longer prior to the first dose of study drug
* is unable or unwilling to discontinue predefined prohibited medications listed in the protocol (refer to section 4.2.3) for 14 days or five half-lives of a drug (whichever is longer) prior to first dose of study drug and for the duration of the study
* any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia
* known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib
* psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol
* clinically assessed as having inadequate venous access for PK sampling
* any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
* legal incapacity or limited legal capacity
* Participation in another clinical study with experimental therapy within the 30 days before start of treatment
* Subjects housed in an institution on official or legal orders
* Pregnancy or lactation period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2012-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Phase I: Assessment of dose-limiting toxicity in order to determine the maximum tolerated dose (MTD) of pazopanib in combination with weekly topotecan | after 4 weeks
  Dose-limiting toxicities are defined as follows:
  * grade 3 or 4 non-hematologic toxicity other than nausea or vomiting
  * grade 3 or 4 thrombocytopenia (platelet count less than 50000/µl)
  * grade 4 neutropenia lasting ≥ 7 days or febrile neutropenia defined as ANC <1000/µl concurrent with fever
  * Any grade 2 and more toxicity of cycle 1 other than nausea, vomiting, rash, alopecia or anemia, that persisted over 35 days.
• Phase II: Progression-free survival according to RECIST criteria | up to 3.5 years
  • Phase II: Progression-free survival according to RECIST criteria

SECONDARY OUTCOMES:
• Overall survival | up to 3.5 years
  • Overall survival
• Response rate (CR, PR) according to RECIST criteria | up to 3.5 years
  • Response rate (CR, PR) according to RECIST criteria
• Clinical benefit rate (CR, PR, SD) | up to 3.5 years
  • Clinical benefit rate (CR, PR, SD)
• Duration of response | up to 3.5 years
  • Duration of response
• Time to progression (TTP) | up to 3.5 years
  • Time to progression (TTP)
• Evaluation of CA-125 tumour response | up to 3.5 years
  • Evaluation of CA-125 tumour response
Safety and tolerability of pazopanib in combination with weekly topotecan | up to 3.5 years
  Incidence and type of AE in terms of:
  * All AE,
  * Related AE,
  * SAE,
  * Related SAE,
  * NCI-CTC (version 4.0) grade 3 and 4 AE,
  * Related NCI-CTC (version 4.0) grade 3 and 4 AE,
  * AE leading to treatment discontinuation,
  * Incidence of, and reason for, deaths.
• Quality of life as defined by EORTC-QLQ C 30 and Ovar 28 questionnaire | up to 3.5 years
  • Quality of life as defined by EORTC-QLQ C 30 and Ovar 28 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: jalid Sehouli, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Campus Virchow-Klinikum, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chekerov R, Arndt T, Pietzner K, Canzler U, Wimberger P, Strauss HG, Mahner S, Woelber L, de Gregorio N, Stocker G, von Abel E, Neunhoeffer T, Belau AK, Mustea A, Yalinkaya I, Braicu EI, Richter R, Sehouli J; NOGGO ovarian cancer study group. Pazopanib with Topotecan weekly for patients with platinum-resistant or intermediate-sensitive recurrent ovarian cancer: results of a multicentre, open label phase I/II study (TOPAZ). J Cancer Res Clin Oncol. 2023 Aug;149(10):7637-7649. doi: 10.1007/s00432-023-04647-9. Epub 2023 Mar 31. PMID 37000264